CLINICAL TRIAL: NCT06439641
Title: Prevalence and Factors Associated With Sleep Disorders in Inflammatory Bowel Disease: a Cross-sectional Study at Reims University Hospital
Brief Title: Prevalence and Factors Associated With Sleep Disorders in Inflammatory Bowel Disease
Acronym: SOMMICI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PO24032*
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Sleep Disorder
Keywords: Inflammatory Bowel Diseases; Crohn's Disease; Ulcerative Colitis; Sleep Disorders
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Inflammatory bowel diseases (Other): patients with IBD
  Interventions: Other: Ulcerative colitis Disease Activity Index

INTERVENTIONS:
Other: Ulcerative colitis Disease Activity Index — QUESTIONNAIRE - Score between 0 to 12, the higher is the worse

SUMMARY:
Inflammatory bowel diseases (IBD) including Crohn's disease (CD) and ulcerative colitis (UC), are an inflammatory disease that can affect the entire digestive tract from the mouth to the anus for CD and the entire colon and rectum for UC. They mainly affect adolescents and young adults. These pathologies evolve in relapses interspersed with phases of remission. Sometimes associated with extraintestinal manifestations (joint, dermatological, ophthalmological or biliary systems), chronic inflammation of the digestive tract and the resulting symptoms (abdominal pain, diarrhea, rectal syndrome, etc.) lead to a significant alteration in the quality of life of patients in all spheres of activity (professional, sexual, social).

Sleep is a basic neurophysiological state, the normal total duration of which in humans is between six and ten hours per day. It is an essential element of the circadian rhythm in humans, influencing certain cellular functions and in particular the synthesis of cytokines and pro-inflammatory molecules. Sleep disturbances and disruption of the circadian rhythm lead to metabolic and immunological dysfunctions, which may be involved in chronic inflammatory conditions through changes in the immune response.

In the field of IBD, many studies suggest poor sleep quality in patients with IBD. While there seems to be a link between sleep disorders and impaired quality of life with a socio-professional impact in these patients, the links between IBD activity, its treatment and sleep disorders are poorly studied, with discordant results in previous studies.

In order to enrich our knowledge on this topic, the investigators wish to study the prevalence and risk factors associated with sleep disorders in IBD patients in order to improve patients' quality of life

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Crohn's disease (CD) or ulcerative colitis (UC) presenting for consultation or hospitalization in Gastroenterology unit

Exclusion Criteria:

* Patients with an identified sleep pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2024-07-03 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index Questionnaire | Only one time at inclusion
  Score between 0 to 12, the higher is the worse

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: No